CLINICAL TRIAL: NCT00916760
Title: Clinical, Multi-centre, Randomised, Double-blind Placebo-controlled Subcutaneous Immunotherapy Trial With Depigmented, Polymerized Extract of Parietaria Judaica Pollen on Patients With Hypersensitivity to This Pollen
Brief Title: Subcutaneous Immunotherapy Treatment for Patients With Hypersensitivity to Parietaria Judaica
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-005871-17
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2012-08

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: allergic, rhinoconjunctivitis, Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): A Subcutaneous Depigmented and Polymerized Allergen extract of Parietaria Judaica 1000 DPP/ml. Depigoid Parietaria judaica 1000 DPP/ml.
  Interventions: Biological: Depigoid Parietaria judaica 1000DPP/ml
- 2 (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Depigoid Parietaria judaica 1000DPP/ml — Subcutaneous monthly treatment
  Other Names: A suspension of depigmented and glutaraldehyde-polymerised allergen extract of Parietaria judaica adsorbed onto aluminium hydroxide.
  Arms: 1
Biological: Placebo — Subcutaneous monthly treatment
  Arms: 2

SUMMARY:
The objective of this trial is to assess the clinical efficacy of the modified extract (depigmented and polymerized with glutaraldehyde) of the subcutaneous injection of Parietaria Judaica pollen in the treatment of patients affected by allergic rhinitis/rhinoconjunctivitis ( with or without episodic asthma) induced by hypersensitivity to grass pollen, evaluating the score regarding symptoms and consumption of the medication.

DETAILED DESCRIPTION:
Immunotherapy is a specific treatment for allergic diseases. Unlike conventional pharmacological treatment, immunotherapy is the only treatment that could modify the natural course of allergic disease. This is a prospective double-blind placebo controlled study with two arms of treatment: placebo and active.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent, signed by the subject
* Positive clinical history of rhinitis/rhinoconjunctivitis allergy to Parietaria pollen
* Patient of both gender aged from 18 up to 55
* Diagnosed Sensitivity to Parietaria pollen base on:

Positive Nasal provocation test Positive prick test to P. Judaica Specific IgE to P.Judaica >0,7KU/L

- Patients who are able to comply with the dose regime

Exclusion Criteria:

* Relevant sensitivity to another perenne allergen
* Patient with asthma
* Use of immunotherapy during the last four years
* Treatment with B. Blocking agents
* Patient suffering from some pathology in which adrenaline was contraindicated
* Subject suffers from a serious medical condition, which would interference the treatment and follow up of the subject in the study
* Subject suffers from autoimmune disease(thyroiditis, lupus, etc.)
* Conditions in which the patient can not offer full co-operation nad significant psychiatric disturbance.
* Intolerance to aspirin
* Pregnant women or with pregnancy risk and brest-feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2008-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Symptoms score | 2 years

SECONDARY OUTCOMES:
Nasal Provocation test, Dose- response skin prick test, Quality of life questionnaire, visual scales, asthma symptom scores, Medication scores, adverse event and severity adverse event,unplanned healthcare resource utilization | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Angel Ferrer, Dr, Principal Investigator — Hospital Vega Baja
Locations (11):
- Spain (11):
  - H. Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Viladecans, Barcelona, Barcelona
  - Hospital Vega Baja, Alicante, Orihuela
  - H. de sagunto, Sagunto, Sagunto
  - Hospital General de Onteniente, Ontinyent, Valencia
  - Hospital Luis Alcañiz, Xàtiva, Valencia
  - Hospital Marina Baixa, Alicante
  - Hospital de Castellón, Castellon
  - Hospital Reina Sofía, Murcia
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital La Fe, Valencia